CLINICAL TRIAL: NCT00350077
Title: The Effect of High Dose Versus Low Dose Intravenous Vitamin C (Ascorbic Acid)on Burn Injury Resuscitation
Brief Title: The Effect of High Dose Vitamin C in Burn Patients
Acronym: Vitamin C
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate resources to submit for approval
Sponsor: United States Army Institute of Surgical Research (U.S. Federal Agency)
Collaborators: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-05-045
Record Dates: First submitted 2006-07-06; First posted 2006-07-10 (Estimated); Last update posted 2011-12-20 (Estimated); Status verified 2011-12

CONDITIONS: Burns
Keywords: Burns
MeSH Terms: conditions — Burns | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Intravenous Vitamin C — vitamin C IV during 24 hour period following burn
Drug: Vitamin C — IV vitamin C

SUMMARY:
The purpose of this study is to see if intravenous Vitamin C will decrease the amount of IV fluids needed following burn injury in the first 48 hours.

DETAILED DESCRIPTION:
Adequate fluid resuscitation in burn injured patients to allow adequate renal blood flow has been the hallmark of burn care in the last 50 years. The danger of exceeding the optimal intravenous fluid resuscitation has resulted in severe complications including abdominal compartment syndrome, loss of upper airway control, extremity compartment syndromes and pulmonary edema. Hig dose vitamin C infusion during the first 24 hours of burn resuscitation has been documented to decrease the overall amount of intravenous fluid needed to provide for adequate renal perfusion and hemodynamic stability in multiple animal model studies. High dose vitamin C is thought to decrease postburn microvascular protein and fluid leakage by reducing postburn lipid oxygenation caused by burn injury generated free radicals.

ELIGIBILITY:
Inclusion Criteria:

* >/= 20% total body surface area full and partial thickness burns
* Admitted to the USAISR burn center within 10 hours post injury

Exclusion Criteria:

* Pregnant or breast feeding
* Documented preadmission or admission renal failure
* History of glucose-6-phosphate dehydrogenase deficiency, kidney stoves, gout or sickle cell
* Electrical injury
* Renal replacement of any kind<24 hours after admission

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-07; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Document a significantly lower intravenous fluid requirement per percent total body surface area burn in the High Dose Vitamin C group | 72 hours
Document a significantly higher number of mechanical ventilator free days | 7 days
Document a significantly lower complication and infection rate in the Vitamin C group | 7 days
Document decreased lipid peroxidation by monitoring serum malondialdehyde (MDA) level | 72 hours

SECONDARY OUTCOMES:
Document a lower incidence of organ failure | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Lorne H Blackbourne, MD, Principal Investigator — United States Army Institute of Surgical Research
Locations (1):
- United States Army Institute of Surgical Research, Fort Sam Houston, Texas, United States

REFERENCES:
- [Background] Matsuda T, Tanaka H, Yuasa H, Forrest R, Matsuda H, Hanumadass M, Reyes H. The effects of high-dose vitamin C therapy on postburn lipid peroxidation. J Burn Care Rehabil. 1993 Nov-Dec;14(6):624-9. doi: 10.1097/00004630-199311000-00007. PMID 8300697
- [Background] Tanaka H, Matsuda T, Miyagantani Y, Yukioka T, Matsuda H, Shimazaki S. Reduction of resuscitation fluid volumes in severely burned patients using ascorbic acid administration: a randomized, prospective study. Arch Surg. 2000 Mar;135(3):326-31. doi: 10.1001/archsurg.135.3.326. PMID 10722036